CLINICAL TRIAL: NCT04631289
Title: Association of Preadmission Metformin Exposure and Incidence of Acute Kidney Injury Within 7 Days in Patients With Type 2 Diabetes in Intensive Care Unit: a Retrospective Cohort Study
Brief Title: Preadmission Metformin Exposure and Incidence of Acute Kidney Injury
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: met on AKI
Record Dates: First submitted 2020-11-12; First posted 2020-11-17 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: AKI
Keywords: Metformin;AKI; Type 2 diabetes; ICU
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- metformin/non-metformin group: Preadmission metformin exposure was defined as a record of metformin usage in "Medications on admission" in MIMIC-III.
  Metformin group included non-AKI type 2 diabetes patients with preadmission metformin exposure.
  Non-metformin group included non-AKI type 2 diabetes patients without preadmission metformin exposure.

SUMMARY:
More than 50% of ICU patients suffer from Acute kidney injury (AKI). Metformin shows protective properties in kidney disease. Our study aimed to validate AKI incidence among diabetes patients in the ICU with or without preadmission metformin exposure. We included non-AKI patients with type 2 diabetes in Medical Information Mart for Intensive Care (MIMIC)-III database. Incidence of AKI and mortality were compared between those with and without preadmission prescriptions.

DETAILED DESCRIPTION:
Emerged as a major public healthy problem, Acute kidney injury (AKI) is now influencing millions of people worldwide and leading to reduced survival, increased progression of latent chronic kidney disease (CKD), and even new onset of CKD. More than half of intensive care unit (ICU) patients underwent AKI in a recent multinational cross-sectional study, often resulting in the need for renal replacement therapy with a high socio-economic impact for the patients.The effective precaution and treatment strategy remains limited.

As the most general and first-line biguanide antihyperglycemic drug, metformin has anti-inflammatory characteristics and is related with decreased all-cause mortality compared with other antihyperglycemics.. In some clinical trials and experimental studies conducted on divergent rodent models representing various types of kidney diseases going from AKI to CKD, metformin has been shown beneficial effects on the kidney. Moreover, preadmission metformin exposure is associated with a lower rate of 28-day mortality among AKI patients showed in several clinical studies.

However, in critical care patients with type 2 diabetes, the evidence of preadmission metformin usage decreasing a risk of AKI incidence is still absented. Therefore we performed a retrospective cohort study to validate the association of preadmission metformin exposure and AKI incidence in patients with diabetes in the ICU .

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes
* >16 years old and <90 years old
* without AKI

Exclusion Criteria:

* CKD
* data error
* type 1 diabetes
* diabetes patients with pregnancy
* no metformin record
* with AKI

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Type 2 diabetes patients without AKI were eligible in our study. AKI was defined according to the Kidney Disease: Improving Global Outcomes (KDIGO) criteria. KDIGO criteria are as follows: increase in SCr to ≥1.5 times baseline must have occurred within the prior 7 days; or ≥0.3 mg/dl increase in serum creatinine (SCr) occurred within 48 h; or urine volume <0.5 ml/kg/h for 6 h or more. The minimum of the SCr values available within the 7 days before admission was used as the baseline SCr[12]. When the preadmission SCr was not available, the first SCr measured at admission was used as the baseline SCr. The diagnosis of type 2 diabetes was based on International Classification of Disease, Ninth Revision (ICD-9). We only included adult patients (age>16 years).
Sampling Method: Probability Sample
Enrollment: 3841 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-11-10 (Actual)

PRIMARY OUTCOMES:
Incidence of AKI | within 7days in the ICU
  AKI was defined according to the Kidney Disease: Improving Global Outcomes (KDIGO) criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Shikun Qian, Principal Investigator — Second Affiliated Hospital of Guangzhou Medical University
Locations (1):
- SAHGuangzhouMU, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided